CLINICAL TRIAL: NCT04310150
Title: Collagen-thrombin Matrix Efficacy During Cardiac Surgery: a Prospective Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2017-0094
Record Dates: First submitted 2020-03-12; First posted 2020-03-17 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Coronary Artery Disease
Keywords: Bleeding; Blood transfusion; Coronary artery bypass surgery; Hemostasis; Topical therapy
MeSH Terms: conditions — Coronary Artery Disease; Hemorrhage | interventions — Collagen

STUDY DESIGN:
Intervention Model Description: In cardiac surgery, patients were randomized to receive Floseal® or Collastat® (n=40), respectively. The selected agent was applied in the operating room.
Who Masked: Participant
Masking Description: The agent was selected using the sealed envelope system. The selected agent was prepared immediately prior to use after randomization, and was delivered to the site of bleeding via a single-barrel syringe.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment arm label- Collastat® (Experimental)
  Interventions: Drug: Collastat
- Control arm label- Floseal® (Active Comparator): an marketed product is Floseal
  Interventions: Device: Floseal

INTERVENTIONS:
Drug: Collastat — hemostatic agent that combine porcine-derived collagen thrombin
  Other Names: absorbable collagen hemostasis
  Arms: Treatment arm label- Collastat®
Device: Floseal — hemostatic agent that combine bovine-derived gelatin
  Other Names: absorbable collagen hemostasis
  Arms: Control arm label- Floseal®

SUMMARY:
In this prospective open-label randomized trial, 160 patients with elective off-pump coronary artery bypass (OPCAB) surgery were enrolled. After primary suture of aortocoronary anastomosis, if an area of hemorrhage was identified, patients were randomized to receive Floseal® or Collastat® (n=80), respectively. The selected agent was applied with compression of the target area for 1 min. If hemostasis was not achieved, the agent was re-applied for a further 1 min, and was repeated up to 5 min, after which rescue treatment was applied, including any conventional surgical methods.

DETAILED DESCRIPTION:
[Patients] A total of 160 patients were enrolled over a 24-month period in a prospective randomized controlled trial between March 2018 and Feburary 2020. The Institutional Review Board (IRB) at our site approved the study prior to patient enrollment (Severance Hospital, South Korea, IRB number; 1-2017-0094), and the study was performed in accordance with the ethical standards as laid down in the 1964 Declaration of Helsinki and its later amendments. Informed consent was obtained prior to the operative procedure. The inclusion criteria for enrollment eligibility specified patients aged 19 years or older, undergoing elective OPCAB surgery with multi-vessel coronary artery disease. Patients were excluded if they were pregnant or had a known sensitivity to any components of the bovine thrombin preparations or the porcine or bovine origin materials. The patients who were taking antithrombotic or antiplatelet agents for more than one week, except for aspirin, or who had hematologic disease were also excluded from this study.

[Procedure and scoring system according to hemostatic status] Baseline complete blood count with differential, activated partial thromboplastin time (aPTT), prothrombin time, electrolyte, and hepatic or renal panel were drawn within 24 hours prior to surgery. Patient enrollment occurred in the operating room when an aortocoronary bypass was finally determined. After full median sternotomy, heparin (0.7-1.0 mg/kg) was administered to achieve the target activated clotting time (ACT; >300 sec). In all patients, a saphenous vein or radial artery grafts were anastomosed to the aorta using the Heartstring device (MAQUET Holding B.V. & Co. KG, Rastatt, Germany). After identification of an aortocoronary anastomosis site, patients were offered the allocated treatment regimen for one of the 2 hemostatic agents, Floseal® or Collastat®, using the sealed envelope system. The selected agent was prepared immediately prior to use after randomization, and was delivered to the site of bleeding via a single-barrel syringe, and light compression was applied with a wet gauze until the bleeding stopped.

We defined the scoring system according to hemostasis status including the following details. At first, the bleeding site was characterized as oozing or pulsatile. The hemostasis status was graded using the 3 steps method (0: no bleeding, 1: oozing, and 2: active bleeding). The treatment was applied with pressure to the target area for 1 min. If hemostasis was achieved within this time, the time to hemostasis was recorded as 1 min. If hemostasis was not achieved, the treatment was re-applied for a further 1 min. if hemostasis was not achieved after 5 min, conventional surgical suture was performed.

Protamine was administered at the end of the OPCAB procedure. The pericardium was loosely closed after the surgery, the midline sternotomy was closed in layers, and 2 mediastinal drains were left in place. Participants in both groups took aspirin 100 mg and clopidogrel 75 mg daily from the first postoperative day. Patients with hemoglobin (Hb) values below 60 g/L always received transfusion therapy. In stable patients with Hb values between 60 and 100 g/L, an evaluation of the patients' clinical status was necessary to determine if transfusion is warranted (Grade of recommendation: 1C+). Transfusion of fresh frozen plasma (FFP) was indicated for the following: correction of congenital deficiencies of clotting factors for which a specific concentrate did not exist; for multiple acquired deficiencies; when the prothrombin time or aPTT, expressed as a ratio, was greater than 1.5; microvascular bleeding in patients undergoing massive transfusion; acute disseminated intravascular coagulation in the presence of ongoing bleeding; together with correction of the underlying cause (Grade of recommendation: 1C+). The platelet concentrates were indicated if the count was below 50x109/L and there was ongoing excessive bleeding (Grade of recommendation: 2C).

[Definition of terms and Endpoint] The following definition was used for application of the agents in the clinical setting: successful hemostasis was achieved when there was cessation of visible bleeding after completion of the hemostatic agent administration.

The primary end points were the proportion of patients with complete hemostasis within 5 min for the aortocoronary anastomosis site treated by hemostatic agents Floseal® or Collastat® and the proportion of patients with complete hemostasis evaluated at 1, 2, and every minute up to 5 minutes. Secondary end points were the time required for hemostasis, blood loss in the operative day, amount of blood products transfused both intraoperatively and postoperatively, rate of surgical revision for bleeding, total length of intensive care unit (ICU) stay, and rate of postoperative morbidity/ mortality.

ELIGIBILITY:
Inclusion Criteria:

1. patients aged 19 years or older
2. undergoing elective OPCAB surgery with multi-vessel coronary artery disease.

Exclusion Criteria:

1. patients were pregnant
2. had a known sensitivity to any components of the bovine thrombin preparations or the porcine origin materials.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with complete hemostasis | Participants will be followed for the time required for hemostasis, an expected average of 3 minutes.
  The primary end points were the proportion of patients with complete hemostasis within or up to 5 min for the aortocoronary anastomosis site treated by hemostatic agents Floseal® or Collastat®

SECONDARY OUTCOMES:
blood loss in the operative day | 24 hours later after surgery
amount of blood products transfused both intraoperatively and postoperatively | 24 hours later after surgery
rate of surgical revision for bleeding | 5 minutes later after anastomosis
total length of intensive care unit (ICU) stay | mean 3-4 days after surgery
rate of postoperative morbidity/mortality | Participants will be followed during 1 years from operation

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee H, Lee JH, Jeon CS, Ko JH, Park SN, Lee YT. Evaluation of a novel collagen hemostatic matrix in a porcine heart and cardiac vessel injury model. J Thorac Dis. 2019 Jul;11(7):2722-2729. doi: 10.21037/jtd.2019.06.59. PMID 31463099
- [Derived] Kim HH, Lee KJ, Kang DR, Lee JH, Youn YN. Hemostatic efficacy of a flowable collagen-thrombin matrix during coronary artery bypass grafting: a double-blind randomized controlled trial. J Cardiothorac Surg. 2023 Jun 15;18(1):193. doi: 10.1186/s13019-023-02196-3. PMID 37322537
- See also: Collastat absorbable collagen hemostatic agent, which provides effective hemostasis for bleeding in high-pressure great vessel. — http://www.dalimmedical.co.kr/board/bbs/board.php?bo_table=product&wr_id=80&sct=new&sct2=